CLINICAL TRIAL: NCT04732663
Title: Understanding Exertional Dyspnea and Exercise Intolerance in COVID-19
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00107436
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Covid19; Dyspnea
Keywords: DLCO; Pulmonary Capillary Blood Volume; VO2peak; Exercise Capacity; Cardiac Function; Impedance Cardiography; Echocardiography; Shortness of Breath; Ventilatory Efficiency; Lung Restriction
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Persistently Symptomatic Covid-19 (PS-CoV): PS-CoV will be defined as individuals with a history of molecular testing confirmed COVID-19 infection, recovered from acute infection but with ongoing symptoms (self-reported, pulmonary, cardiac, musculoskeletal or other symptoms) of at least 4 weeks' duration. Recovery from acute infection will be defined according to provincial health guidelines: at least 10 days' (14 in those hospitalized; 21 in those with immunocompromise) from onset of symptoms with at least 24 hours without a fever, without taking anti-pyretic medications and improvement of other symptoms.
  Interventions: Other: No Intervention
- Recovered Covid-19: Recovered Covid-19 Survivors will be defined as individuals without complaint of a persisting covid-19 symptom. Recovered Covid-19 survivors will be matched to PS-CoV for age, sex, body mass index and time post corona virus infection.
  Interventions: Other: No Intervention
- Control: Covid Naïve Controls will be defined as individuals who have no known history of covid-19. Control participants will be matched to PS-CoV for age, sex and body mass index.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Cross-sectional study, no intervention.

SUMMARY:
A novel corona virus emerged in 2019 causing Corona Virus Disease 2019 (covid-19). In one year more than 80 000 000 cases worldwide were documented. Some patients experience symptoms, specifically shortness of breath, long after the viral infection has passed. These patients are colloquially known as "Covid-19 Long-Haulers" and it is currently unknown why symptoms remain after infection.

Shortness of breath and exercise intolerance may be caused by corona virus infection, covid-19 therapy, and reduced physical activity. Exercise intolerance may be due to lung, heart, blood vessel and muscle changes. During infection, the corona virus appears to cause lung blood vessel and gas exchange surface damage. Early reports show heart dysfunction, secondary to pulmonary blood vessel dysfunction or damage. Critically, no data is available on lung blood vessel function or cardiac function during exercise. Moreover, no data are available to link persistent symptoms to physiology parameters. To better understand symptom persistence in Covid-19, the investigators aim to measure exercise tolerance and heart and lung function in covid-19 survivors and compare them to covid-19 free controls.

DETAILED DESCRIPTION:
Purpose and Justification:

In less than one year, the novel coronavirus has infected more than 80 000 000 people worldwide. Infection causes Corona Virus Disease 2019 (covid-19) and in some cases severe acute respiratory syndrome. Overall risk of mortality from covid-19 is low, however, risk radically increases with age and cardiovascular comorbidity. The long-term consequences of covid-19 are not known. Already a phenotype of survivors with prolonged symptom burden has presented; this phenotype is characterized by persistent respiratory (cough, sputum, dyspnea, wheeze) and musculoskeletal (pain, fatigue) symptoms. Preliminary data from clinical exercise testing conducted at the UofA pulmonary function laboratory suggests covid-19 survivors with prolonged symptoms have significantly reduced exercise tolerance and increased exertional dyspnea.

Impaired exercise tolerance measured as peak oxygen uptake (VO2peak) is the strongest independent predictor of cardiovascular and all-cause mortality. The investigators preliminary data in seven persistently symptomatic covid-19 survivors (PS-CoV) 3-months post molecular confirmation of infection shows a mean 30% impairment in VO2peak relative to age-, sex- and body mass index matched controls. Several facets of covid-19, including treatment and recovery, may contribute to the range and severity of debilitation and impairment in VO2peak in PS-CoV. The purpose of this study is to investigate impairments in VO2peak, and pulmonary, cardiac and peripheral factors contributing to impaired VO2peak, exercise intolerance, and persistent dyspnea in PS-CoV.

Coronavirus gains cellular entry through binding angiotensin converting enzyme in the lungs, making the lungs and pulmonary vasculature a logical starting point for investigation of persistent symptomology. During active infection, pulmonary vascular dysfunction, microthromboemboli, micro-angiopathy and pulmonary inflammation and/or fibrosis are reported. Accompanying this is a reduction in diffusion capacity at rest, increased tortuosity of pulmonary vasculature, and elevated pulmonary vascular resistance. One mechanistic explanation is that regions downstream of micro-thromboemboli become fibrotic secondary to reduced blood flow resulting in reduced diffusion capacity. Physiological adaptation through intussusceptive angiogenesis results in increased tortuosity of pulmonary vasculature, with a secondary consequence of increased pulmonary vascular resistance. However, evidence of isolated decreases in diffusion capacity in the absence of pulmonary fibrosis are at odds with this theory. An alternative explanation is that pulmonary vascular dysfunction precedes lesions viewed by computed tomography (CT) and changes in lung volumes. Regardless of incipient damage, for ~1/3 of hospitalized covid-19 patients, the end result is pulmonary fibrosis, impaired diffusion capacity (measured as the diffusion limitation of carbon monoxide, DLCO), reduced forced vital capacity (FVC) and proportionately reduced forced expiratory volume in one second (FEV1).

In PS-CoV, lung impairment at 3-month follow-up is characterized by reduced resting DLCO, FVC and FEV1, and incomplete normalization of pulmonary CT consolidation and opacities.13 The investigators preliminary data in PS-CoV show increased respiratory rate and VE/VCO2 (indicative of increased deadspace or excessive ventilatory drive) at peak exercise- characteristic of parenchymal or restrictive lung disease and consistent with pathology of covid-19 including parenchymal cell death and pulmonary fibrosis. Despite these findings, initial data suggest that PS-CoV patients' operating lung volumes during exercise and peak breathing reserve are relatively preserved. Previous work in COPD has shown that an elevated VE/VCO2 during exercise is explained by higher deadspace, and this increased VE/VCO2 contributes to increased dyspnea secondary to increased drive to breathe. The investigators work in COPD has shown that the increase VE/VCO2 is due to hypoperfusion of the pulmonary capillaries as demonstrated by a reduced DLCO and reduced pulmonary capillary blood volume during exercise, and that when pulmonary perfusion is improved by using inspired NO, VE/VCO2 and dyspnea are decreased resulting in an increase in VO2peak.

No data are currently available examining symptoms of dyspnea, pulmonary mechanics, VE/VCO2, and impaired VO2peak in PS-CoV. Moreover, no data are available examining diffusion capacity or pulmonary capillary blood volume responses during exercise, which may contribute to increased VE/VCO2, pulmonary inefficiency, perceived dyspnea, and secondary cardiac consequences.

Cardiac complications of covid-19 have been demonstrated and may contribute to impaired VO2peak through a reduction in peak cardiac output (Qpeak). Limited data are available, but, cardiac effects appear to be (mal)adaptation secondary to pulmonary vascular dysfunction, angiopathy and increased pulmonary vascular resistance. Importantly, pulmonary vascular dysfunction may impose a cardiac limitation to exercise in the absence of or preceding structural cardiac changes as in early pulmonary hypertension (exercise induced pulmonary hypertension). Complications mimic those observed in pulmonary hypertension whereby the thin walled right ventricle insidiously adapts to and eventually fails against chronically increased pulmonary artery pressure. This includes right ventricular hypertrophy, dilation and hypokinesis, and in failure, uncoupling of tricuspid annular plane systolic excursion (TAPSE) and pulmonary artery systolic pressure (PASP). In a study of 100 consecutive covid-19 patients at rest, 39% of patients had right ventricular dilation and dysfunction and 16% of patients had left ventricular diastolic dysfunction. No reports of cardiac function during exercise or cardiac mechanics in response to stress are available following covid-19, and it is unknown whether cardiac consequences of covid-19 limit VO2peak or contribute to symptom persistence in PS-CoV.

Detrimental changes in body composition occur in hospitalized covid-19 patients. During active infection, frailty (in part characterized by muscle loss) is associated with increased covid-19 severity and mortality. Reduced lean tissue mass and increased adiposity, particularly in the thigh, are reported following bedrest and are known to impair VO2peak. Reductions in VO2peak are twofold: absolute VO2peak is reduced due to loss of muscle mass, and relative VO2peak (ml/kg/min) is reduced due to a combination of reduced absolute VO2peak and a decrease in the ratio of muscle mass to total body mass. Moreover, bedrest is associated with reduced mitochondrial density and oxidative enzymatic activity. No data are available linking increased adiposity, reduced thigh muscle, or impaired muscle quality to VO2peak or symptom persistence in PS-CoV.

The investigators preliminary data indicate VO2peak is impaired in PS-CoV survivors. The magnitude of VO2peak, pulmonary, cardiac and peripheral impairment is not known in PS-CoV or symptom free covid-19 survivors. Through this proposed study, the investigators aim to comprehensively test VO2peak impairment in PS-CoV survivors and link physiology to symptom persistence in covid-19.

Objectives:

There are 3 objectives of this study: 1) to evaluate VO2peak in PS-CoV and recovered covid-19 survivors (no longer symptomatic) compared to covid-19 naïve controls matched for age, sex and body mass index; 2) to evaluate DLCO and pulmonary capillary blood volume at rest and during exercise in these three groups; and 3) evaluate cardiac structure and function at rest and during exercise in the three groups.

Hypotheses:

The investigators hypothesize that:

1. VO2peak will be impaired in PS-CoV relative to recovered (symptom free) covid-19 survivors and covid naïve controls, and that recovered covid-19 survivors will have impaired VO2peak relative to covid naïve controls;
2. Relative to covid-19 naïve controls, PS-CoV will have reduced rest and exercise pulmonary capillary blood volume and diffusion capacity, which will be correlated with exercise VE/VCO2.
3. PS-CoV will have reduced peak cardiac output, increased PASP, and uncoupling of PASP:TAPSE.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19/Symptom status as defined under each group.

Exclusion Criteria:

1. Previous diagnosis of pulmonary hypertension
2. Obesity (body mass index >30 kg/m2)
3. Absolute contraindication to exercise testing or an orthopedic limitation that may interfere with cardiopulmonary exercise testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with or without a history of covid-19, with or without persistent symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Peak Oxygen Uptake (VO2peak) | Within 20-30 seconds of completion of trial
  Staged cardiopulmonary exercise test
Peak Cardiac Output (Qpeak) | Within 20-30 seconds of completion of trial
  Impedance cardiography derived Qpeak from staged CPET
Pulmonary Capillary Blood Volume (Vc) | Averaged across trials
  Multiple fraction of inspired oxygen DLCO derived pulmonary capillary blood volume at rest and during exercise.

SECONDARY OUTCOMES:
Ventilatory Efficiency (VE/VCO2) | Averaged across trial
  Measured from expired gas analysis during cardiopulmonary exercise testing.
Dyspnea | Assessed every 2-minutes until completion of the exercise trial; anticipating ~10-14 minute tests
  Measured using the modified Borg scale (1-10, 10=maximal dyspnea), perceived dyspnea during cardiopulmonary exercise testing.
  Scale = 1-10
Membrane Diffusion Capacity (Dm) | Averaged across trials
  Measured at rest and during exercise using the multiple fraction of inspired oxygen DLCO technique.
Pulmonary Artery Systolic Pressure (PASP) | Assessed for five consecutive cardiac cycles and are measured in triplicate during the cardiac ultrasound trial
  Echocardiography estimated pulmonary artery systolic pressure.
Right Ventricular Function | Assessed for five consecutive cardiac cycles and are measured in triplicate during the cardiac ultrasound trial
  Reported as PASP:TAPSE (tricuspid annular plane systolic excursion) measured using echocardiography.
Left Ventricular Stiffness | Assessed for five consecutive cardiac cycles and are measured in triplicate during the cardiac ultrasound trial
  Estimated from E/e' using echocardiography.

OTHER OUTCOMES:
Physical Activity | Step count averaged across 5 days
  Self reported physical activity and accelerometer based physical activity monitoring (Fitbit).
Thigh Composition | Assessed at rest and are measured in triplicate
  Muscle and adipose thickness, muscle echo intensity (ultrasound).
Frailty | Assessed upon admission
  Questionnaire assessment (Edmonton Frail Scale, FRAIL Scale, Frailty Phenotype, or Clinical Frail Scale)
Quality of Life (QoL) | Assessed upon admission
  Health related quality of life as assessed using the Post Covid Functional Scale, EQ5D-5L
Hemoglobin | Pre and post exercise trial
  Blood hemoglobin concentration (finger prick)
Muscle Oxygenation | Assessed at rest and are measured in triplicate
  Quadriceps muscle oxygenation during exercise measured by near infrared spectroscopy.
Blood Biomarkers | Assessed upon admission
  Biomarkers of inflammation, organ and tissue damage including CRP, INFg, BNP, CK.

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, Ph.D., Principal Investigator — University of Alberta
Locations (1):
- Clinical Physiology Laboratory, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanyaolu A, Okorie C, Marinkovic A, Patidar R, Younis K, Desai P, Hosein Z, Padda I, Mangat J, Altaf M. Comorbidity and its Impact on Patients with COVID-19. SN Compr Clin Med. 2020;2(8):1069-1076. doi: 10.1007/s42399-020-00363-4. Epub 2020 Jun 25. PMID 32838147
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Myers J, Prakash M, Froelicher V, Do D, Partington S, Atwood JE. Exercise capacity and mortality among men referred for exercise testing. N Engl J Med. 2002 Mar 14;346(11):793-801. doi: 10.1056/NEJMoa011858. PMID 11893790
- [Background] Quinn KL, Fralick M, Zipursky JS, Stall NM. Renin-angiotensin-aldosterone system inhibitors and COVID-19. CMAJ. 2020 May 19;192(20):E553-E554. doi: 10.1503/cmaj.200619. Epub 2020 Apr 24. No abstract available. PMID 32332039
- [Background] Malas MB, Naazie IN, Elsayed N, Mathlouthi A, Marmor R, Clary B. Thromboembolism risk of COVID-19 is high and associated with a higher risk of mortality: A systematic review and meta-analysis. EClinicalMedicine. 2020 Dec;29:100639. doi: 10.1016/j.eclinm.2020.100639. Epub 2020 Nov 20. PMID 33251499
- [Background] Zhao YM, Shang YM, Song WB, Li QQ, Xie H, Xu QF, Jia JL, Li LM, Mao HL, Zhou XM, Luo H, Gao YF, Xu AG. Follow-up study of the pulmonary function and related physiological characteristics of COVID-19 survivors three months after recovery. EClinicalMedicine. 2020 Aug;25:100463. doi: 10.1016/j.eclinm.2020.100463. Epub 2020 Jul 15. PMID 32838236
- [Background] Dhawan RT, Gopalan D, Howard L, Vicente A, Park M, Manalan K, Wallner I, Marsden P, Dave S, Branley H, Russell G, Dharmarajah N, Kon OM. Beyond the clot: perfusion imaging of the pulmonary vasculature after COVID-19. Lancet Respir Med. 2021 Jan;9(1):107-116. doi: 10.1016/S2213-2600(20)30407-0. Epub 2020 Nov 17. PMID 33217366
- [Background] Merrill JT, Erkan D, Winakur J, James JA. Emerging evidence of a COVID-19 thrombotic syndrome has treatment implications. Nat Rev Rheumatol. 2020 Oct;16(10):581-589. doi: 10.1038/s41584-020-0474-5. Epub 2020 Jul 30. PMID 32733003
- [Background] Huang Y, Tan C, Wu J, Chen M, Wang Z, Luo L, Zhou X, Liu X, Huang X, Yuan S, Chen C, Gao F, Huang J, Shan H, Liu J. Impact of coronavirus disease 2019 on pulmonary function in early convalescence phase. Respir Res. 2020 Jun 29;21(1):163. doi: 10.1186/s12931-020-01429-6. PMID 32600344
- [Background] Lang M, Som A, Carey D, Reid N, Mendoza DP, Flores EJ, Li MD, Shepard JO, Little BP. Pulmonary Vascular Manifestations of COVID-19 Pneumonia. Radiol Cardiothorac Imaging. 2020 Jun 18;2(3):e200277. doi: 10.1148/ryct.2020200277. eCollection 2020 Jun. PMID 34036264
- [Background] Ackermann M, Mentzer SJ, Kolb M, Jonigk D. Inflammation and intussusceptive angiogenesis in COVID-19: everything in and out of flow. Eur Respir J. 2020 Nov 12;56(5):2003147. doi: 10.1183/13993003.03147-2020. Print 2020 Nov. PMID 33008942
- [Background] Burel-Vandenbos F, Cardot-Leccia N, Passeron T. Pulmonary Vascular Pathology in Covid-19. N Engl J Med. 2020 Aug 27;383(9):886-887. doi: 10.1056/NEJMc2022068. Epub 2020 Jul 17. No abstract available. PMID 32678531
- [Background] Sonnweber T, Sahanic S, Pizzini A, Luger A, Schwabl C, Sonnweber B, Kurz K, Koppelstatter S, Haschka D, Petzer V, Boehm A, Aichner M, Tymoszuk P, Lener D, Theurl M, Lorsbach-Kohler A, Tancevski A, Schapfl A, Schaber M, Hilbe R, Nairz M, Puchner B, Huttenberger D, Tschurtschenthaler C, Asshoff M, Peer A, Hartig F, Bellmann R, Joannidis M, Gollmann-Tepekoylu C, Holfeld J, Feuchtner G, Egger A, Hoermann G, Schroll A, Fritsche G, Wildner S, Bellmann-Weiler R, Kirchmair R, Helbok R, Prosch H, Rieder D, Trajanoski Z, Kronenberg F, Woll E, Weiss G, Widmann G, Loffler-Ragg J, Tancevski I. Cardiopulmonary recovery after COVID-19: an observational prospective multicentre trial. Eur Respir J. 2021 Apr 29;57(4):2003481. doi: 10.1183/13993003.03481-2020. Print 2021 Apr. PMID 33303539
- [Background] Tedjasaputra V, Bouwsema MM, Stickland MK. Effect of aerobic fitness on capillary blood volume and diffusing membrane capacity responses to exercise. J Physiol. 2016 Aug 1;594(15):4359-70. doi: 10.1113/JP272037. Epub 2016 May 12. PMID 26959808
- [Background] Tedjasaputra V, van Diepen S, Phillips DB, Wong EYL, Bhutani M, Michaelchuk WW, Bryan TL, Stickland MK. Pulmonary capillary blood volume response to exercise is diminished in mild chronic obstructive pulmonary disease. Respir Med. 2018 Dec;145:57-65. doi: 10.1016/j.rmed.2018.10.015. Epub 2018 Oct 19. PMID 30509717
- [Background] Szekely Y, Lichter Y, Taieb P, Banai A, Hochstadt A, Merdler I, Gal Oz A, Rothschild E, Baruch G, Peri Y, Arbel Y, Topilsky Y. Spectrum of Cardiac Manifestations in COVID-19: A Systematic Echocardiographic Study. Circulation. 2020 Jul 28;142(4):342-353. doi: 10.1161/CIRCULATIONAHA.120.047971. Epub 2020 May 29. PMID 32469253
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Li Y, Li H, Zhu S, Xie Y, Wang B, He L, Zhang D, Zhang Y, Yuan H, Wu C, Sun W, Zhang Y, Li M, Cui L, Cai Y, Wang J, Yang Y, Lv Q, Zhang L, Xie M. Prognostic Value of Right Ventricular Longitudinal Strain in Patients With COVID-19. JACC Cardiovasc Imaging. 2020 Nov;13(11):2287-2299. doi: 10.1016/j.jcmg.2020.04.014. Epub 2020 Apr 28. PMID 32654963
- [Background] Oliveira RKF, Faria-Urbina M, Maron BA, Santos M, Waxman AB, Systrom DM. Functional impact of exercise pulmonary hypertension in patients with borderline resting pulmonary arterial pressure. Pulm Circ. 2017 Jul-Sep;7(3):654-665. doi: 10.1177/2045893217709025. Epub 2017 Jun 8. PMID 28895507
- [Background] Vonk Noordegraaf A, Galie N. The role of the right ventricle in pulmonary arterial hypertension. Eur Respir Rev. 2011 Dec;20(122):243-53. doi: 10.1183/09059180.00006511. PMID 22130817
- [Background] D'Alto M, Marra AM, Severino S, Salzano A, Romeo E, De Rosa R, Stagnaro FM, Pagnano G, Verde R, Murino P, Farro A, Ciccarelli G, Vargas M, Fiorentino G, Servillo G, Gentile I, Corcione A, Cittadini A, Naeije R, Golino P. Right ventricular-arterial uncoupling independently predicts survival in COVID-19 ARDS. Crit Care. 2020 Nov 30;24(1):670. doi: 10.1186/s13054-020-03385-5. PMID 33256813
- [Background] Gualtieri P, Falcone C, Romano L, Macheda S, Correale P, Arciello P, Polimeni N, Lorenzo A. Body Composition Findings by Computed Tomography in SARS-CoV-2 Patients: Increased Risk of Muscle Wasting in Obesity. Int J Mol Sci. 2020 Jun 30;21(13):4670. doi: 10.3390/ijms21134670. PMID 32630032
- [Background] Hewitt J, Carter B, Vilches-Moraga A, Quinn TJ, Braude P, Verduri A, Pearce L, Stechman M, Short R, Price A, Collins JT, Bruce E, Einarsson A, Rickard F, Mitchell E, Holloway M, Hesford J, Barlow-Pay F, Clini E, Myint PK, Moug SJ, McCarthy K; COPE Study Collaborators. The effect of frailty on survival in patients with COVID-19 (COPE): a multicentre, European, observational cohort study. Lancet Public Health. 2020 Aug;5(8):e444-e451. doi: 10.1016/S2468-2667(20)30146-8. Epub 2020 Jun 30. PMID 32619408
- [Background] Ma Y, Hou L, Yang X, Huang Z, Yang X, Zhao N, He M, Shi Y, Kang Y, Yue J, Wu C. The association between frailty and severe disease among COVID-19 patients aged over 60 years in China: a prospective cohort study. BMC Med. 2020 Sep 7;18(1):274. doi: 10.1186/s12916-020-01761-0. PMID 32892742
- [Background] McGuire DK, Levine BD, Williamson JW, Snell PG, Blomqvist CG, Saltin B, Mitchell JH. A 30-year follow-up of the Dallas Bedrest and Training Study: II. Effect of age on cardiovascular adaptation to exercise training. Circulation. 2001 Sep 18;104(12):1358-66. PMID 11560850
- [Background] Ferretti G, Antonutto G, Denis C, Hoppeler H, Minetti AE, Narici MV, Desplanches D. The interplay of central and peripheral factors in limiting maximal O2 consumption in man after prolonged bed rest. J Physiol. 1997 Jun 15;501 ( Pt 3)(Pt 3):677-86. doi: 10.1111/j.1469-7793.1997.677bm.x. PMID 9218227